CLINICAL TRIAL: NCT06931132
Title: Cancer-related Fatigue and Symptom Clusters - Effects of Virtual, Imagined and Real-life Nature-based Therapy in Cancer Survivors - a RCT
Brief Title: Cancer-related Fatigue and Symptom Clusters - Effects of Virtual, Imagined and Real-life Nature-based Therapy in Cancer Survivors
Acronym: FOREST
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Robert Bosch Gesellschaft für Medizinische Forschung mbH (RBMF) (Other)
Collaborators: Wuerzburg University Hospital (Other); University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Marcela Winkler, MD, Head of Integrative Medicine, Robert Bosch Gesellschaft für Medizinische Forschung mbH (RBMF)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: S00855-NIM
Record Dates: First submitted 2025-04-01; First posted 2025-04-17 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-04

CONDITIONS: Cancer Survivors
Keywords: Fatigue; Forest therapie; Virtual Reality
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Real-life FOREST bathing (Experimental)
  Interventions: Other: Real-life forest bathing
- Simulated FOREST bathing (Virtual Reality). (Experimental)
  Interventions: Other: Simulated FOREST bathing (Virtual Reality)
- Imaging FOREST bathing. (Experimental)
  Interventions: Other: Imaging FOREST bathing
- Wait-list group (No Intervention)

INTERVENTIONS:
Other: Real-life forest bathing — Participants will experience the elements (olfactory, acoustic and haptic) of forest bathing for 30 minutes (sitting) in a forested area. The forests have been previously selected near Stuttgart and Würzburg and are comparable to each other.
  Arms: Real-life FOREST bathing
Other: Simulated FOREST bathing (Virtual Reality) — Using virtual reality goggles, a FOREST bathing experience will be simulated. The simulation will have elements of the classic FOREST bathing (olfatory, acoustic and haptic) and will last 30 minutes.
  Arms: Simulated FOREST bathing (Virtual Reality).
Other: Imaging FOREST bathing — A therapist will lead an imaginative exercise in which participants will imagine a FOREST bathing. The imaginative exercise will include elements of the classic FOREST bathing (olfactory, acoustic and haptic) and will last 30 minutes.
  Arms: Imaging FOREST bathing.

SUMMARY:
This is a randomized, controlled, bicenter trial comparing the effects on symptoms and quality of life in cancer survivors. Three nature-based therapies will be compared with a wait-list group. The therapies are: virtual reality simulated forest, guided imaging and classic forest bathing. Each intervention lasts 30 minutes and takes place once a week for 8 weeks. All interventions involve different stimulus types: visual, olfactory, auditory and tactile.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have completed treatment for cancer (*with the exception of long-term adjuvant endocrine therapy).
* Subjective Impairment due to Cancer-Related Fatigue (CrF) . NCCN-recommended questions are used for screening ("How exhausted do you feel on a scale of 0 to 10?" and "How impaired do you feel by this fatigue on a scale of 0 to 10?" (threshold >4 on either scale).
* At the time of study inclusion, it must be expected that no further antitumor therapy measures will be started within the next 6 months.
* Patients must be able to refrain from smoking up to 15 minutes before the intervention (smoking within 15 minutes before therapy impairs the participant's ability to perceive the aroma of the phytoncides).
* Written and valid informed consent from the patient.

Exclusion Criteria:

* Presence of inadequately controlled major depression in the opinion of the investigator.
* Asthma (inhaled phytoncides may cause airway irritation, exacerbation of asthma, or bronchoconstriction).
* Known allergy to pine or citrus fragrance.
* Anosmie.
* Medical history of seasickness (virtual reality can cause nausea/vomiting with no improvement after 5-10 minutes).
* History of seizures (virtual reality may increase susceptibility to seizures due to the changing light in the forest video).
* Visual and hearing impairments that are not corrected by visual or hearing aids.
* Unwillingness to store and share personal medical data as part of the protocol.
* Participation in another clinical trial focusing on behavioural or complementary medicine interventions.
* Missing or incomplete consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Fatigue | 8 weeks (end of intervention)
  The Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) is a validated tool for the reliable measurement of fatigue in patients with cancer and other chronic diseases. The questionnaire has high internal consistency and validity and allows assessment of fatigue and its impact on quality of life and disease progression. 13 items to measure self-reported fatigue and its impact on daily activities and functions. Scores range from 0 to 52, with higher scores indicating less fatigue (better outcome).
Sleep | 8 weeks (end of intervention)
  The Pittsburgh Sleep Quality Index (PSQI) measures subjective sleep quality. The 19-item questionnaire generates seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medications, and daytime disturbances. The sum of the scores for these seven components gives a global score. Scores range from 0 to 21, with higher scores indicating poorer sleep quality (worse outcome).
Depression | 8 weeks (end of intervention)
  The Patient Health Questionnaire-9 (PHQ-9) is often used for the initial diagnosis of depression and for monitoring the course of the illness. The PHQ-9 consists of 9 questions that ask about the main and core symptoms of depression over the past two weeks, providing a structured and objective assessment of the severity of depression. Scores range from 0 to 27, with higher scores indicating more severe depression (worse outcome).
Concentration | 8 weeks (end of intervention)
  The Functional Assessment of Cancer Therapy - Cognitive Function (FACT-Cog) is a 5-point Likert scale measure of chemotherapy-induced cognitive impairment in cancer patients. The questionnaire consists of 24 items covering four different domains: self-perceived cognitive impairment, feedback from others, perceived cognitive ability, and impact on quality of life. The assessment of these cognitive aspects indicates a relationship with objective symptoms and allows for a nuanced assessment of treatment-induced cognitive impairment. Scores range from 0 to 148, with higher scores indicating better perceived cognitive functioning (better outcome).

SECONDARY OUTCOMES:
Fatigue | 8 weeks (end of intervention)
  The Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) is a validated tool for the reliable measurement of fatigue in patients with cancer and other chronic diseases. The questionnaire has high internal consistency and validity and allows assessment of fatigue and its impact on quality of life and disease progression. 13 items to measure self-reported fatigue and its impact on daily activities and functions. In addition to the primary outcome (overall fatigue score), this secondary outcome will focus on specific FACIT-F items related to fatigue interference in daily activities. This aims to explore functional limitations due to fatigue beyond the global score. Scores range from 0 to 52, with higher scores indicating less fatigue (better outcome).
Sleep | 8 weeks (end of intervention)
  The Pittsburgh Sleep Quality Index (PSQI) measures subjective sleep quality. The 19-item questionnaire generates seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medications, and daytime disturbances. The sum of the scores for these seven components gives a global score. Scores range from 0 to 21, with higher scores indicating worse sleep quality (worse outcome).
Depression | 8 weeks (end of intervention)
  The Patient Health Questionnaire-9 (PHQ-9) is often used for the initial diagnosis of depression and for monitoring the course of the illness. The PHQ-9 consists of 9 questions that ask about the main and core symptoms of depression over the past two weeks, providing a structured and objective assessment of the severity of depression. Scores range from 0 to 27, with higher scores indicating more severe depressive symptoms (worse outcome).
Concentration | 8 weeks (End of intervention)
  The Functional Assessment of Cancer Therapy - Cognitive Function (FACT-Cog) is a 5-point Likert scale measure of chemotherapy-induced cognitive impairment in cancer patients. The questionnaire consists of 24 items covering four different domains: self-perceived cognitive impairment, feedback from others, perceived cognitive ability, and impact on quality of life. The assessment of these cognitive aspects indicates a relationship with objective symptoms and allows for a nuanced assessment of treatment-induced cognitive impairment. Scores range from 0 to 148, with higher scores indicating better cognitive function (better outcome).
Resilience | 8 weeks (end of intervention)
  The Brief Resilience Scale (BRS) is a instrument used to measure resilience, or an individual's ability to bounce back quickly from stress, adversity, or challenge. The BRS is known for its brevity and conciseness, with only a few items rated on a Likert scale. Scores range from 1 to 5, with higher scores indicating greater resilience (better outcome).
Mindfulness | 8 weeks (end of intervention)
  The Mindfulness Awareness Scale (MAAS) measures a person's level of mindfulness. The scale ranges from 1 to 6 and includes a total of 15 items. The items assess the extent to which a person invests his or her thoughts in the present moment by taking into account the extent to which he or she is aware of what is going on in his or her environment at any given moment. Scores range from 15 to 90, with higher scores indicating greater mindfulness (better outcome).
Anxiety | 8 weeks (end of intervention)
  The Generalized Anxiety Disorder-7 (GAD-7) is a standardized screening questionnaire used to assess the severity of generalized anxiety disorder. It is used in both clinical practice and research to rapidly identify and assess the severity of anxiety symptoms. The questionnaire consists of 7 items that ask about typical symptoms of generalized anxiety disorder and focus on the last two weeks. Scores range from 0 to 21, with higher scores indicating more severe anxiety (worse outcome)
Quality of life Questionnaire | 8 weeks (end of intervention)
  Functional Assessment of Cancer Therapy - (FACT-G) Quality of Life Questionnaire. The FACT-G was developed through a structured process to identify relevant content for a cancer-specific quality of life questionnaire. The instrument allows the calculation of a generic total quality of life scale (FACT-G) as well as subscales for physical, social, emotional, and functional quality of life. Scores range from 0 to 108, with higher scores indicating better quality of life (better outcome).
Sensation of stress | 8 weeks (end of intervention)
  The Perceived Stress Scale (PSS) is the most frequently used psychological instrument for measuring the perception of stress. It measures the degree to which situations in a person's life are perceived as stressful. The scale also includes a series of direct questions about the current experience of stress. The items are easy to understand and the response alternatives are easy to record. The questionnaire consists of 10 items. Scores range from 0 to 40, with higher scores indicating greater perceived stress (worse outcome).
Simulator Disease (Virtual reality group only, arm 2) | 8 weeks (end of intervention)
  The Simulator Sickness Questionnaire (SSQ) is a standardised instrument designed to assess symptoms of simulator or motion sickness commonly experienced when using virtual reality (VR) and other simulated environments. The instrument consists of a series of questions divided into three subscales: Nausea, Disorientation and Oculomotor Stress.
  The SSQ is widely used in VR research as it provides a means of quantifying symptoms and assessing their severity. Studies have shown that the SSQ is valid and reliable and has a high correlation with actual experienced symptoms. The results of the SSQ can be used to optimise VR experiences and improve usability. Total scores range from 0 to 235.62, with higher scores indicating greater simulator sickness (worse outcome).
Physical Activity and Sport Questionnaire | 8 weeks (end of intervention)
  Physical activity will be assessed using the Physical Activity and Sport Questionnaire (BSA), which records the frequency and type of physical activity in the past 4 weeks. Scores will be calculated in MET-minutes/week, based on self-reported duration and intensity of different physical activity domains (work, leisure, sport). Higher scores indicate higher levels of physical activity (better outcome).
Safety evaluation | Through 8 weeks of intervention (Weeks 0-8)
  To assess safety, participants will be asked whether they experienced any adverse events (AEs) during the 8-week intervention period. All reported AEs will be documented and classified by type and severity according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
  The outcome will be the number of participants with at least one treatment-related adverse event recorded from baseline through the end of the 8-week intervention.
Average daily step count (measured via wearable activity tracker) | Cumulative average daily steps over Weeks 1-8
  Physical activity will be monitored continuously during the 8-week intervention using a commercially available wearable device (e.g., Fitbit or Garmin).
  The tracker will record daily step counts, active minutes and movement intensity.
  The outcome will be the average number of steps per day during Week 8, as a marker of overall movement behavior. This complements patient-reported activity recorded in the physical activity diary.
Heart rate variability | 8 weeks (end of intervention)
  Heart Rate Variability (HRV) is measured to assess autonomic nervous system activity and stress recovery. HRV will be recorded using a wearable chest strap sensor (e.g., Polar H10) or equivalent device, over a 5-minute resting period.
  Outcome will be RMSSD (Root Mean Square of Successive Differences) in milliseconds.
Natural killer cell activity | 8 weeks (end of intervention)
  Natural killer (NK) cell activity will be assessed by blood sampling at baseline and Week 8. Cytotoxic activity will be measured by flow cytometry based on CD107a expression and IFN-gamma production.
  Outcome will be the percentage of NK cells expressing CD107a after stimulation.
Serum cytokine concentrations (IL-6, IL-10, TNF-alpha) | Week 4 (Mid-intervention), Week 8 (End of intervention)
  Serum cytokines (IL-6, IL-10, TNF-alpha) will be measured using multiplex ELISA from venous blood samples collected at baseline, Week 4 and Week 8.
  Outcomes will be reported as individual changes in cytokine concentrations (pg/mL) from baseline to Week 4 and Week 8.Outcomes will be reported as individual changes in cytokine concentrations (pg/mL); no composite score will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Loeffler, Dr., Principal Investigator — Würzburg University. Würzburg, Bayern, Germany, 97080; Marcela Winkler, Dr., Principal Investigator — Robert-Bosch-Krankenhaus, Stuttgart, Baden Würtemberg, Germany, 70341
Locations (2):
- Germany (2):
  - Dr med. Marcela Winkler, Stuttgart, Baden-Wurttemberg
  - PD Dr. Claudia Löffler, Würzburg, Bavaria